CLINICAL TRIAL: NCT00827944
Title: ProGrip Mesh Repair Versus Lichtenstein Mesh Repair: a Comparative Randomized Study in Primary Inguinal Hernia
Brief Title: Parietex Progrip Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SC 0607/1
Record Dates: First submitted 2009-01-22; First posted 2009-01-23 (Estimated); Results first posted 2016-11-17 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Hernia, Inguinal
Keywords: Uncomplicated primary inguinal hernias
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Parietex ProGrip
  Interventions: Device: Parietex Progrip
- 2 (Active Comparator): Low weight polypropylene mesh
  Interventions: Device: Low weight polypropylene mesh

INTERVENTIONS:
Device: Parietex Progrip — Surgical technique:
  Self-gripping lightweight Polyester and Polylactic acid meshes providing a sutureless fixation.
  Arms: 1
Device: Low weight polypropylene mesh — Surgical technique:
  Lichtenstein repair with lightweight polypropylene mesh (inferior to 70gr/m2) secured to the posterior inguinal wall with sutures
  Arms: 2

SUMMARY:
The objective of the study is to evaluate pain and disabling complications inducing social consequences in primary inguinal hernia ProGrip mesh repair compared to Lichtenstein repair with lightweight polypropylene mesh.

DETAILED DESCRIPTION:
* Patients in ProGrip group will be treated with self-gripping lightweight Polyester and Polylactic acid meshes providing a sutureless fixation.
* Patients in Lichtenstein group will be treated with lightweight Polypropylene meshes requiring fixation by sutures.
* Study participation will start at signature of informed consent and each patient will be assessed before surgery. A close follow-up will be performed: 7 days (questionnaires and phone call), 1 month (clinical visit), 3 months (questionnaires and phone call), and final evaluation at 12 months (clinical visit) after surgery, which will end the participation to the study.
* 600 adult males divided in 2 groups requiring primary uncomplicated elective inguinal hernia mesh repair will be included in the study. Patients will be stratified by center.

ELIGIBILITY:
Inclusion Criteria:

* All male patients at participating centers with a primary, uncomplicated inguinal hernia.
* Collar of the defect ≤ 4 cm
* Signed informed consent

Exclusion Criteria:

* 30 years ≥ Age ≥ 75 years
* Emergency procedure
* Inclusion in other trials
* Bilateral inguinal hernia
* Recurrence

Ages: 31 Years to 74 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 603 (Actual)
Dates: Start 2008-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- Universitaire Ziekenhuizen Leuven, Leuven, Belgium
- Germany (2):
  - Klinikum Bremen-Mitte, Bremen
  - Herz-Jesu-Krankenhaus gGmbH, Chirurgische Klinik, Fulda
- Catharina-ziekenhuis, Eindhoven, Netherlands
- Sweden (2):
  - Medical Center Linköping, Linköping
  - Centre of clinical research, Västeras-
- United Kingdom (3):
  - Western Infirmary, Glasgow
  - Imperial College London / Faculty of Medecine, London
  - Derriford Hospital, Plymouth

REFERENCES:
- [Derived] Sanders DL, Nienhuijs S, Ziprin P, Miserez M, Gingell-Littlejohn M, Smeds S. Randomized clinical trial comparing self-gripping mesh with suture fixation of lightweight polypropylene mesh in open inguinal hernia repair. Br J Surg. 2014 Oct;101(11):1373-82; discussion 1382. doi: 10.1002/bjs.9598. Epub 2014 Aug 21. PMID 25146918

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study period: 42 months First patient in: 13 October 2008 Last patient in: 27 April 2011 Last Patient visit: 8 May 2012 Follow-up duration: 1 year
Groups:
- Progrip Group: Parietex ProGrip
  Parietex Progrip : Surgical technique:
  Self-gripping lightweight Polyester and Polylactic acid meshes providing a sutureless fixation.
- Lichtenstein Group: Low weight polypropylene mesh
  Low weight polypropylene mesh : Surgical technique:
  Lichtenstein repair with lightweight polypropylene mesh (inferior to 70gr/m2) secured to the posterior inguinal wall with sutures
Period: Overall Study
Arm/Group | Progrip Group | Lichtenstein Group
Started | 304 | 299
Completed | 241 | 240
Not Completed | 63 | 59

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Progrip Group | Lichtenstein Group | Total
Number analyzed (Participants) | 304 | 299 | 603
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (12.1) | 57.2 (10.9) | 57.2 (11.5)
Gender [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 304 | 299 | 603
Region of Enrollment [Number; unit: participants]
  Belgium | 13 | 12 | 25
  Germany | 54 | 53 | 107
  Netherlands | 58 | 59 | 117
  United Kingdom | 92 | 89 | 181
  Sweden | 87 | 86 | 173

OUTCOME MEASURES:

1. Secondary Outcome: Foreign Body Sensation
Description: Foreign body sensation using a specific questionnaire at M1, M3, M12 months after surgery. Questionnaire will be completed by patient during consultation or will be sent to the patient with instructions to complete it and send it back by mailing.
Time Frame: M1, M3, M12 months after surgery
Population: The analysis were performed on an As Treated population, with a 5% significance level.
Measure: Number; unit: participants
Arm/Group | Progrip Group | Lichtenstein Group
Number analyzed (Participants) | 304 | 299
participants
  FBS at Rest - M1 (Answer : No) | 159 | 173
  FBS Normal Activities - M1 (Answer: No) | 139 | 148
  FBS Doing exercise - M1 (Answer : No) | 121 | 128
  FBS General Feeling - M1 (Answer : No) | 144 | 151
  FBS at Rest - M3 (Answer : No) | 186 | 198
  FBS Normal Activities - M3 (Answer: No) | 166 | 177
  FBS Doing exercise - M3 (Answer : No) | 140 | 155
  FBS General feeling - M3 (Answer : No) | 172 | 189
  FBS at Rest - M12 (Answer : No) | 178 | 196
  FBS Normal Activities - M12 (Answer: No) | 169 | 197
  FBS Doing exercise - M12 (Answer : No) | 171 | 165
  FBS General Feeling - M12 (Answer : No) | 176 | 199

2. Secondary Outcome: Chronic Pain Defined as Pain Lasting More Than 3 Months Using VAS Score
Description: Chronic pain defined as pain lasting more than 3 months using VAS score. A VAS going from 0 mm (no pain) to 150 mm (worst conceivable pain) is presented to the patient who draw a vertical line on the scale to indicate the average amount of pain at the time of consultation or at home.
Time Frame: 3 months after surgery
Measure: Number; unit: participants
Arm/Group | Progrip Group | Lichtenstein Group
Number analyzed (Participants) | 241 | 240
participants | 9 | 12

3. Primary Outcome: Pain Assessment During the First Three Months and at One Year After Surgery Using a Visual Analogue Scale (VAS)
Description: Pain assessment during patient follow up after surgery using VAS score. VAS going from 0 mm (no pain) to 150 mm (worst conceivable pain) is presented to the patient who draw a vertical line on the scale to indicate the average amount of pain at the time of consultation or at home.
Time Frame: M3, M12 after surgery
Population: The analysis were performed on an As Treated (AT)population, with a 5% significance level.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Progrip Group | Lichtenstein Group
Number analyzed (Participants) | 241 | 240
units on a scale
  VAS - 3 months | 7.48 (15.82) | 6.76 (17.05)
  VAS - 12 months | 4.62 (10.81) | 5.27 (13.27)

4. Primary Outcome: Pain Assessment During the First Three Months and at One Year After Surgery Using a Surgical Pain Scales (SPS)
Description: Surgical pain scales (=SPS) completed by patient during consultation or will be sent to the patient with instructions to complete it and send it back by mailing. The score of evaluation will be reported in mm, specifying if pain occurs at rest, during normal activities, during exercise. The score is ranged from 0 (no pain) to 150 mm (the worst pain yu have never known).
Time Frame: M3, M12 after surgery
Population: The analysis were performed on an As Treated population (AT), with a 5% significance level.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Progrip Group | Lichtenstein Group
Number analyzed (Participants) | 241 | 240
units on a scale
  Surgical Pain - 3 months | 6.62 (15.42) | 7.85 (15.52)
  Surgical Pain - 12 months | 5.51 (15.12) | 4.37 (9.77)

5. Secondary Outcome: Wound Complications and Hernia Recurrences
Time Frame: M12 after surgery
Population: The analysis were performed on an As Treated (AT) population, with a 5% significance level.
Measure: Number; unit: participants
Arm/Group | Progrip Group | Lichtenstein Group
Number analyzed (Participants) | 262 | 267
participants
  Seroma | 4 | 6
  Hematoma | 13 | 5
  Site Surgical Infection | 9 | 14
  Recurrence | 4 | 8

6. Secondary Outcome: Return to Work and to Normal Daily Activities
Time Frame: Effective date
Population: The analysis were performed on an As Treated (AT) population, with a 5% significance level.
Measure: Mean (Standard Error); unit: days
Arm/Group | Progrip Group | Lichtenstein Group
Number analyzed (Participants) | 304 | 299
days
  Return to work | 14.61 (11.61) | 14.79 (11.51)
  Return to daily activities | 7.99 (8.78) | 8.426 (8.145)

7. Secondary Outcome: Other Post-operative Complications
Time Frame: M12 after surgery
Population: As Treated population
Measure: Number; unit: participants
Arm/Group | Progrip Group | Lichtenstein Group
Number analyzed (Participants) | 262 | 267
participants | 23 | 29

ADVERSE EVENTS:
Time Frame: 12 months after surgery
Groups:
- Progrip Group: Parietex ProGrip
  Surgical technique: Self-gripping lightweight Polyester and Polylactic acid meshes providing a sutureless fixation.
- Lichtenstein Group: Low weight polypropylene mesh
  Surgical technique: Lichtenstein repair with lightweight polypropylene mesh (inferior to 70gr/m2) secured to the posterior inguinal wall with sutures
Arm/Group | Progrip Group | Lichtenstein Group
Serious Adverse Events (participants affected / at risk) | 18/304 | 21/299
Other Adverse Events (participants affected / at risk) | 23/304 | 29/299
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Progrip Group (N=304) | Lichtenstein Group (N=299)
Ischemic left testis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
High pain just after surgery, ilioinguinal nerve trapped in suture (General disorders) | 0 (0) | 1 (1)
Inguinal hernia recurrence (Surgical and medical procedures) | 4 (4) | 5 (5)
Right Total Hip Replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
inguinal pain after lifting a heavy weight, suspected hernia recurrence (General disorders) | 0 (0) | 1 (1)
Acute retention of urine (Renal and urinary disorders) | 1 (1) | 0 (0)
prostate adenocarcinoma (Renal and urinary disorders) | 1 (1) | 0 (0)
Hand Tendon Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ureter transection left, direct suture (Renal and urinary disorders) | 1 (1) | 0 (0)
Melena red blood loss per anum Hospitalisation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pulmonary sarcoïdosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
atrial flutter (Vascular disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Vascular disorders) | 0 (0) | 1 (1)
lungmetastasis dorsolateral right lung (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
necrotic defect 0,5cm scar pace maker (Cardiac disorders) | 1 (1) | 0 (0)
Lung Embol (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Elective trans-urethral resection of prostate (Reproductive system and breast disorders) | 0 (0) | 1 (1)
edema, poor kidney function, decompensation cordes, pneumonia (General disorders) | 0 (0) | 1 (1)
enlarged prostate gland resulting in surgical intervention (Reproductive system and breast disorders) | 1 (1) | 0 (0)
HERNIA RECURRENCE ADMISSION FOR REPAIR (Surgical and medical procedures) | 0 (0) | 1 (1)
NEURALGIC PAIN RIGHT GROIN (post-op) (General disorders) | 0 (0) | 1 (1)
hospitalization surgery umbilical hernia (Surgical and medical procedures) | 0 (0) | 1 (1)
Cancer colon + metastasis liver and spleen (Gastrointestinal disorders) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Hematoma (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Increasing pain in the inguinal area (General disorders) | 1 (1) | 0 (0)
Gastric Ulcus Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
neuronitis vestibularis left (Eye disorders) | 1 (1) | 0 (0)
acute on chronic renal insufficiency (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Progrip Group (N=304) | Lichtenstein Group (N=299)
Seroma (Skin and subcutaneous tissue disorders) | 4 (4) | 6 (6)
Hematoma (Skin and subcutaneous tissue disorders) | 13 (13) | 5 (5)
Site Surgical Infection (Skin and subcutaneous tissue disorders) | 9 (9) | 14 (14)
Recurrence (Skin and subcutaneous tissue disorders) | 4 (4) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less